CLINICAL TRIAL: NCT00484809
Title: A Post-Marketing Surveillance Looking at Safety of Enbrel (Etanercept) in Adults With Active Rheumatoid Arthritis (RA) and Children With Juvenile Rheumatoid Arthritis (JRA).
Brief Title: Study Evaluating the Tolerance and Safety of Enbrel (Etanercept) in Adults and Children
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0881A-101511
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2007-12-14 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; juvenile rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Juvenile | interventions — Etanercept

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Enbrel (Etanercept)

SUMMARY:
This postmarketing surveillance study will evaluate the safety profile of Enbrel (etanercept) in an Indian population. It will provide surveillance on a currently approved indication for Enbrel of reducing symptoms and inhibiting the progression of structural damage in patients with moderately to severely active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in this study will be as per the approved indications in the package insert.
* Patients with moderately to severely active RA.
* Children with JRA who have had an inadequate response to one or more DMARDs.

Exclusion Criteria:

* Known hypersensitivity to etanercept or any of its components.
* Known significant concurrent medical disease, including:

  * Congestive heart failure, uncontrolled angina pectoris, recent history of myocardial infarction
  * Cancer or history of cancer
  * Active infection
  * Sepsis or risk of sepsis
  * Active tuberculosis or a past history of tuberculosis
  * Pancytopenia
* Females who are pregnant, breast feeding or at risk of pregnancy and not using a medically acceptable form of contraception.
* Patients who are planning to undergo elective surgery during the study period.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2004-03; Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer